CLINICAL TRIAL: NCT02813954
Title: The Predictive Value of Amniotic Fluid pH and Electrolytes on Neonatal Respiratory Disorders
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seda Yilmaz Semerci, Postdoctoral Fellow of Neonatology, MD, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 12
Record Dates: First submitted 2016-06-22; First posted 2016-06-27 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Respiratory Distress Syndrome; Transient Tachypnea of Newborn
MeSH Terms: conditions — Respiratory Distress Syndrome; Transient Tachypnea of the Newborn

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Study Group: Neonates with respiratory distress
  Interventions: Device: Blood Gas Sampling
- Control Group: Healthy Infants

INTERVENTIONS:
Device: Blood Gas Sampling — analyzing amniotic fluid by blood gas device
  Groups: Study Group

SUMMARY:
Amniotic fluid (AF) is a complex structure with a changing content by gestational time. AF pH can be affected by both maternal and fetal conditions such as preterm ruptures of membranes, prematurity and fetal distress. While fetal urine is the major content of AF since 20th gestational week, fetal lung liquid (FLL) also acts as a minor content. Secretion of FLL depends on chloride transport and postnatal clearance of FLL is provided by active reabsorption of sodium (Na) ions. Down-regulation of epithelial Na channels (ENaCs) and an increase of pulmonary compliance accompany to pulmonary adaptation developing at the first hours of life. Lower genomic expression of Na channels in airways is shown to be associated to respiratory distress syndrome (RDS) in preterm. Although pH and electrolyte value of AF is thought to be relevant to fetal and maternal conditions such as gestational age, antenatal steroids and preterm birth, there is no study about this topic in the literature.

ELIGIBILITY:
Inclusion Criteria:

Accepted to participate with informed consent Normal healthy pregnancies

Exclusion Criteria:

Congenital abnormalities Chromosomal abnormalities Blood contaminated AF Declined to participate

Max Age: 25 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 184 (Actual)
Dates: Start 2015-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The Predictive Value of Amniotic Fluid pH and Electrolytes on Neonatal Respiratory Disorders | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Seda Yilmaz Semerci, Principal Investigator — Postdoctoral Fellow of Neonatology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yilmaz Semerci S, Yucel B, Erbas IM, Gunkaya OS, Talmac M, Cetinkaya M. The utility of amniotic fluid pH and electrolytes for prediction of neonatal respiratory disorders. J Matern Fetal Neonatal Med. 2020 Jan;33(2):253-257. doi: 10.1080/14767058.2018.1488961. Epub 2018 Jul 22. PMID 30033781